CLINICAL TRIAL: NCT05546853
Title: Study Investigating the Association of NP137 With mFOLFIRINOX in Locally Advanced Pancreatic Ductal Adenocarcinoma
Acronym: LAP-NET1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: NETRIS Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC22.0211
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — netrin-1 inhibitor NP137; Oxaliplatin; Irinotecan

STUDY DESIGN:
Intervention Model Description: Multicentric prospective single arm phase 1b trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): NP137+ mFOLFIRINOX
  Interventions: Drug: NP137; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Calcium levofolinate; Drug: 5 FU

INTERVENTIONS:
Drug: NP137 — NP137 will be administrated at the first day of each cycle (CnD1) of 14 days as an IV infusion at 9 or 14 mg/kg.
Drug: Oxaliplatin — Oxaliplatin will be administreted at the first day of each cycle (CnD1) of 14 days as an IV infusion at 85 mg/m²
Drug: Irinotecan — Irinotecan will be administreted at the first day of each cycle (CnD1) of 14 days as an IV infusion at 150 mg/m²
Drug: Calcium levofolinate — Calcium levofolinate will be administreted at the first day of each cycle (CnD1) of 14 days as an IV infusion at 100 mg/m²
Drug: 5 FU — 5 FU will be administreted at the first day of each cycle (CnD1) of 14 days as an IV infusion at 2400 mg/m2 as a continuous intravenous infusion over 46 hours.

SUMMARY:
The study will assess the safety of the association of NP137 with the standard of care mFOLFIRINOX in the treatment of locally advanced pancreatic ductal adenocarcinoma.The study drug which is tested is the NP137 in association with mFOLFIRINOX to allow a better tumor response as well as better survival outcomes with an acceptable safety.

DETAILED DESCRIPTION:
The study is a multicentric, prospective, single arm phase 1b trial. This study will enroll 43 to 52 patients and consists of 2 parts: Safety Lead-in Phase and Expansion Phase. Initially, 3 to 12 patients will be enrolled into a Safety Lead-in Phase based on a 3 + 3 design, with the possibility of dose de-escalation, to confirm the recommended dose of NP137.The Expansion Phase will start after completion of Safety Lead-in Phase at the confirmed dose and will include 40 patients. Patients will be assigned to the experimental arm (NP137 + mFOLFIRINOX).

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 79 years
2. Able to understand and sign informed consent
3. Histologically or cytologically proven diagnosis of pancreatic ductal adenocarcinoma
4. Locally advanced pancreatic cancer considered unresectable according to NCCN Guidelines® Version 2.2021
5. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors RECIST 1.1 criteria
6. Male, or non-pregnant and non-lactating female
7. Women patients of childbearing potential* must have a negative serum/urine pregnancy test at screening and baseline, and be willing to use a highly effective** contraception. The patient should be advised to continue the contraception for at least 6 months following the completion of dosing. Women with cessation for > 24 months of previously occurring menses, or women of any age who have had a hysterectomy, or have had both ovaries removed will be considered to be of non-childbearing potential
8. Male patients of reproductive potential must be willing to use one acceptable method of contraception, as judged by Investigator and Sponsor and/or to refrain from donating sperm from the time of screening through at least 6 months following the completion of dose administration
9. No prior systemic therapy, radiation therapy, or resection for pancreatic cancer
10. Life expectancy ≥ 12 weeks
11. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
12. Adequate liver function:

    1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN),
    2. Bilirubin ≤ 1.5 x ULN or in subjects with biliary stenting ≤ 2.0 x ULN
    3. Alkaline phosphatase < 2.5 x ULN
    4. Subjects with biliary stenting do not need to wait for their alkaline phosphatase to become < 2.5 x ULN if their total bilirubin, AST and ALT have improved to within required study levels with criteria 12a and 12b
13. Adequate bone marrow function: platelets >100,000 cells/mm3, hemoglobin > 9.0 g/dl and absolute neutrophil count (ANC) >1,500 cells/mm3
14. Adequate renal function: creatinine < 1.5 x ULN, creatinine clearance ≥ 30 mL/min/m2
15. Adequate nutritional state with Albumin ≥ 2.5 g/dL
16. Less than grade 2 pre-existing peripheral neuropathy (per CTCAE)
17. Patients covered by Health Insurance System

Exclusion Criteria:

1. Patients with resectable pancreatic cancer
2. Evidence of the presence of metastases.
3. Patients who have received prior systemic therapy, radiation therapy, or resection for pancreatic cancer or prior therapy with NP137
4. Patients with known Dihydropyrimidine dehydrogenase (DPD) deficiency, or homozygosity for UGT1A1*28 polymorphism (UGT1A1 genotype analysis is not required to be eligible)
5. Previous (within the past 3 years) or concurrent malignancy diagnosis except non-melanoma skin cancer and in situ carcinomas (excluding in situ breast cancer)
6. History of severe (grade ≥ 3) allergic reactions to one of the components of chemotherapy, or NP137
7. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, may decrease subject's compliance to study's procedures or may render the patient at high risk from treatment complications in the opinion of the treating investigator
8. Subjects with known poorly controlled comorbid conditions, including; congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD), uncontrolled diabetes mellitus (DM) or neurologic disorders (not acutely related to pancreatic cancer) or limited function
9. Major surgery within 4 weeks prior to signing informed consent form. Biliary stents are permitted
10. History of allergy or hypersensitivity to human, humanized or chimeric monoclonal antibodies
11. History of allergy or hypersensitivity to any of the chemotherapy agents belonging to mFOLFIRINOX regimen
12. Subjects with a history of chronic HCV, HBV or HIV infection
13. Subjects who have been administered a live vaccine within four weeks prior to the first administration of therapy
14. Subjects who cannot stop chronic medications that inhibit or induce CYP2C8 or CYP3A4
15. Persons referred to in Articles L1121-5 to L1121-8 of the French code of public health (this corresponds to all persons protected: pregnant or parturient women, breastfeeding mothers, persons deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure)
16. Patients who have active infection requiring systemic therapy (other than HCV, HBV, HIV).
17. Patients who participate or plan to participate in another interventional clinical trial or who is in exclusion period for another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Percentage Proportion of patients experiencing adverse events | At 6 months
  Percentage Proportion of patients experiencing adverse events (AEs) of any grade and grade 3/4 AEs as defined by the National Cancer Institute - Common Terminology Criteria for Adverse Events (CTCAE v 5.0) at 6 months.

SECONDARY OUTCOMES:
Best overall objective response rate (ORR) | At 3,6,9 and 12 months
  Best overall objective response rate (ORR) and ORR at 3 months, 6, 9, 12 months according to RECIST 1.1
Overall survival (OS) | at 6, 12 and 36 months
  Median Overall survival (OS), 6 months and 12 months-OS rates. OS is defined as the time between inclusion and death (all causes). Patients alive will be censored at the date of last news.
Progression-Free Survival (PFS) | at 6, 12 and 36 months
  Median Progression-Free Survival (PFS), 6 months and 12 months-PFS rates. PFS is defined as the time between inclusion and progression according to RECIST 1.1 or death (all causes). Patients alive without progression will be censored at the date of last news.
Median Duration of response | at 6 and 36 months
  Median Duration of response is defined as the time between first dose of treatment and progression according to RECIST 1.1. Patients alive without progression will be censored at 6 months and at the date of last news.
Quality of life (QoL) | at 6 and 36 months
  Quality of life will be studied by using the EORTC QLQ-C30 questionnaire (European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire for Cancer) at 6 months and at the end of study. A 5-point decrease of QLQ-C30 score will be considered as the minimal clinically significant deterioration of QoL.
time to deterioration | at 6 and 36 months
  TTD will be defined as the time from inclusion in the study to deterioration of EORTC QLQ-C30 score with a decrease ≥5 points at any time point after the baseline score, at 6 months and at the end of study
PK-PD evaluation | at 36 months
  PK-PD evaluation: based on available PopPK modelisation and PK samples collected at the time of the response evaluation in this study
CA19.9 response | at 6 and 12 months
  CA19.9 response will be defined as a percentage of patients with a ≥ 50% reduction from baseline CA19.9 level, at 6 and 12 months.
proportion of patients reaching surgery | at 6 and 36 months
  Percentage surgical resection with R0/R1 margins at 6 months and at the end of study.
Mechanisms of EMT | At month 0
  To assess the mechanisms of EMT reversal by comparing different histological markers on pre-therapeutic biopsies with tumor samples obtained during surgical tumor resection. Descriptive study in spatial transcriptomics and immunohistochemistry of the evolution of EMT markers, Netrin-1 expression, and tumor microenvironment by comparing pre-therapeutic biopsies to tumor samples obtained during surgical tumor resection

CONTACTS AND LOCATIONS:
Overall Officials: Gaël ROTH, MD PHD, Principal Investigator — University Hospital, Grenoble
Locations (9):
- France (9):
  - CHU de GRENOBLE ALPES, Grenoble, Alpes
  - CHU de BORDEAUX, Bordeaux, Bordeaux
  - CHU de REIMS, Reims, Reims
  - CHRU Lille, Lille
  - Hôpital Privé Jean Mermoz, Lyon
  - AP-HP Pitié Salpetrière, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU St Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No